CLINICAL TRIAL: NCT00718419
Title: An Open Label, Multicenter Phase 2 Study of Single-Agent Enzastaurin HCl in Previously Treated Waldenstrom's Macroglobulinemia or Multiple Myeloma
Brief Title: A Study for Patients That Have Been Previously Been Treated in Waldenstrom's Macroglobulinemia or Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11481; H6Q-MC-S042 (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Waldenstrom's Macroglobulinemia; Multiple Myeloma
Keywords: Waldenstrom's Macroglobulinemia; Multiple Myeloma
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Multiple Myeloma | interventions — enzastaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A: Enzastaurin (Experimental)
  Interventions: Drug: Enzastaurin

INTERVENTIONS:
Drug: Enzastaurin — Enzastaurin: Cycle 1 Day 1 only: 3, 125-milligrams (mg) tablets three times on Day 1 (Day 1 total dose = 1125 mg)
  Day 2 onwards and subsequent Cycles: 2, 125-mg tablets orally twice a day (500 mg total per day).
  Cycle length (all cycles): 28 days. Patients may stay on drug past 8 cycles, (until the study is closed) or until disease progression.
  Other Names: LY317615

SUMMARY:
To determine whether further study of single-agent enzastaurin is warranted in patients with previously treated Waldenstrom's Macroglobulinemia or Multiple Myeloma based on response.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Patients must have Waldenstrom's Macroglobulinemia (WM) or Multiple Myeloma (MM) previously treated with at least 1 and no more than 5 prior therapies.
* Treatment with prior autologous transplant is permitted. If a transplant is used as consolidation following chemotherapy, without intervening disease progression, it will be considered 1 line of treatment with the preceding chemotherapy.
* Patients with MM must have a monoclonal protein in the serum of greater than or equal to 1 gram per deciliter (g/dL) or monoclonal light chain in the urine protein electrophoresis of greater than or equal to 200 milligrams (mg)/ 24 hours, or measurable plasmacytoma.
* Patients with WM must have an immunoglobulin M (IgM) paraprotein with a minimum IgM level of > 2 times the upper limit of normal (ULN), have detectable lymphoplasmacytic (LPL) cells in the bone marrow, and be symptomatic for WM.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0, 1, or 2.
* The following laboratory values obtained prior to registration:

  * Absolute neutrophil count (ANC) greater than or equal to 1000/microliter
  * Platelet (PLT) count greater than or equal to 75,000/microliter
  * Total bilirubin less than or equal to 1.5 x ULN (if total is elevated check direct and, if normal, patient is eligible)
  * Aspartate transaminase (AST) less than or equal to 3 x ULN
  * Creatinine less than or equal to 1.5 x ULN
  * Hemoglobin (Hgb) greater than or equal to 8.0 g/dL.
* Expected survival of greater than 12 weeks.
* The ability to provide informed consent.
* Male and female patients with reproductive potential must use an approved contraceptive method, if appropriate (for example, intrauterine device [IUD], birth control pills, or barrier device) during and for 3 months after discontinuation of study treatment. Women with childbearing potential must have a negative serum pregnancy test less than or equal to 3 days prior to study enrollment

Exclusion Criteria:

* Prior allogeneic hematopoietic stem cell transplant.
* Are unable to discontinue use of non-Enzyme-Inducing Anti-Epileptic Drugs (EIAEDs), for example carbamazepine, phenobarbital, and phenytoin. Patients on anti-coagulant therapy should be monitored. Ongoing treatment with therapeutic doses of Coumadin is prohibited. However, prophylactic, low dose (less than or equal to 2 mg daily) Coumadin for deep venous thrombosis (DVT) is allowed. In such cases, prothrombin time/ international normalized ratio (PT/INR) should be closely monitored.
* Have electrocardiogram (ECG) abnormalities including baseline 12-lead ECG with QTc interval of greater than 450 milliseconds (msec) in males or greater than 470 msec in females, or QRS duration of greater than 100 msec. Patients who have a congenital long-QT-syndrome in their own or family medical history should be excluded at the investigator's discretion.
* Have an uncontrolled infection.
* Have prior treatment with Carmustine (BCNU) 6 weeks, alkylating agent 4 weeks, or other cytotoxic chemotherapy agents 4 weeks prior to registration in this trial. Have prior treatment with biologic therapy less than or equal to 12 weeks or corticosteroids less than or equal to 2 weeks prior to registration in this trial. However, treatment with less than or equal to 10 mg of prednisone as a chronic therapy is allowed.
* Have radiation therapy less than or equal to 2 weeks prior to treatment in this trial.
* Are pregnant or breast-feeding.
* Are being treated with concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational.
* Are known to be human immunodeficiency virus (HIV) positive.
* Were previously treated with enzastaurin.
* Patients who are unable to swallow tablets.
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Concurrent malignancy that could complicate interpretation of response or safety evaluation. Non-melanoma skin cancer and carcinoma in situ of the cervix are not exclusions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-07; Primary Completion 2010-09 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon- Fri 9 AM- 5 PM Eastern time (UTC/GMT- 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts, United States
- France (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Roche-sur-Yon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nantes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nîmes

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Multiple Myeloma (MM): Participants diagnosed with MM received: Three 125-milligrams (mg) Enzastaurin tablets three times on Day 1 of Cycle 1 (Day 1 total dose = 1125 mg). Day 2 onwards and subsequent Cycles: Two 125-mg tablets orally twice a day (500 mg total per day). Cycle length (all cycles): 28 days.
- Waldenstrom's Macroglobulinemia (WM): Participants diagnosed with WM received: Three 125-milligrams (mg) Enzastaurin tablets three times on Day 1 of Cycle 1 (Day 1 total dose = 1125 mg). Day 2 onwards and subsequent Cycles: Two 125-mg tablets orally twice a day (500 mg total per day). Cycle length (all cycles): 28 days.
Period: Overall Study
Arm/Group | Multiple Myeloma (MM) | Waldenstrom's Macroglobulinemia (WM)
Started | 14 | 42
Received at Least One Dose of Study Drug | 14 | 42
Completed | 1 (Participants who completed 8 cycles of treatment.) | 3 (Participants who completed 8 cycles of treatment.)
Not Completed | 13 | 39
Not completed — Adverse Event | 2 | 1
Not completed — Physician Decision | 1 | 6
Not completed — Sponsor decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 5
Not completed — Progressive Disease | 7 | 25
Not completed — Death Due to Progressive Disease | 2 | 0
Not completed — Death Due to Study Drug Related | 0 | 1
Not completed — Death Due to Adverse Events | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multiple Myeloma (MM) | Waldenstrom's Macroglobulinemia (WM) | Total
Number analyzed (Participants) | 14 | 42 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.28 (7.51) | 64.57 (8.53) | 66.7 (9.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 8 | 35 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African | 0 | 1 | 1
  Caucasian | 14 | 41 | 55
Region of Enrollment [Count of Participants; unit: Participants]
  France | 14 | 5 | 19
  United States | 0 | 37 | 37

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response (CR), Partial Response (PR) and Minimal Response (MR) or Minor Response (MinR): (Response Rate)
Description: European Group for Blood and Bone Marrow Transplant (EBMT) Response Criteria (RC) used for MM. CR: no serum/urine M protein for 6 weeks (wk), <5% plasma cells in bone marrow (PCBM), no lytic bone lesions (LBL) size/number increase, no soft tissue plasmacytomas (STPC); PR: met some CR criteria plus maintain for 6 wk ≥50% serum monoclonal paraprotein (SPEP) and PCBM decrease, either decrease of ≥90% or <200 mg light chain excretion (LCE), ≥50% STPC size decrease; MR: met some PR criteria plus maintain for 6 wk, a decrease of: 25-49% SPEP, 50-89% 24 hour urinary LCE, 25-49% PCBM, 25-49% STPC size. International Workshop on WM (IWWM) RC used for WM. CR: no serum M protein, malignant cells in BM, or lymphadenopathy/organomegaly; PR: ≥50% immunoglobulin M (IgM) and adenopathy/organomegaly (A/O) decrease; no new symptoms of WM. MinR: ≥25% to <50% IgM decrease, no A/O progression; no cytopenias or clinical symptoms of WM.
Time Frame: Baseline to measured progressive disease up to 40.51 months
Population: All participants who received at least one dose of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Multiple Myeloma (MM) | Waldenstrom's Macroglobulinemia (WM)
Number analyzed (Participants) | 14 | 42
percentage of participants | 7.1 | 38.1

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as elapsed time from the first evidence of CR, PR, MR or MinR until date of progression of disease (PD). EBMT RC used for MM. CR: no serum/urine M protein for 6 wk, <5% PCBM, no LBL size/number increase, no STPC; PR: met some CR criteria plus maintain for 6 wk ≥50% SPEP and PCBM decrease, either decrease of ≥90% or <200 mg LCE, ≥50% STPC size decrease; MR: met some PR criteria plus maintain for 6 wk decrease of: 25-49% SPEP, 50-89% 24 hour urinary LCE, 25-49% PCBM, 25-49% STPC size. PD: >25% increase in SPEP, 24 hour urinary LCE, PCBM, STPC size increase, new bone lesion or STPC. IWWM RC used for WM. CR: no serum M protein, malignant cells in BM, or lymphadenopathy/organomegaly; PR: ≥50% IgM and A/O decrease; no new WM symptoms. MinR: ≥25% to <50% IgM decrease, no A/O progression; no cytopenias or clinical of WM symptoms. PD: >25% IgM increase, progression of clinical findings or symptoms. For participants who had no PD, DOR was censored at their last contact.
Time Frame: Time of response to time of measured progressive disease up to 38.37 months
Population: All participants who received at least one dose of the study drug and had complete response (CR) or partial response (PR) or minimal response (MR) or minor response (MinR). The numbers of participants censored are 1 (MM) and 13 (WM).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Multiple Myeloma (MM) | Waldenstrom's Macroglobulinemia (WM)
Number analyzed (Participants) | 1 | 16
months | NA [NA to NA] — Only 1 participant had response, therefore median and 95% Confidence Interval were not calculable. | NA [17.87 to NA] — Only 3 participants had events, therefore median was not calculated. The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

3. Secondary Outcome: Time to Progressive Disease
Description: Time to progression is defined as the elapsed time from the date of study enrollment to the date of objectively determined progressive disease (PD). European Group for Blood and Bone Marrow Transplant (EBMT) Response Criteria was used for MM. PD: >25% increase in serum monoclonal paraprotein (SPEP), 24 hour urinary light chain excretion (LCE), plasma cells in bone marrow (PCBM), soft tissue plasmacytomas (STPC) size increase, new bone lesion or STPC. International Workshop on WM (IWWM) Response Criteria was used for WM. PD: >25% immunoglobulin M (IgM) increase, progression of clinical findings or symptoms. For participants who had no PD, time to PD was censored at their last contact.
Time Frame: Baseline to measured progressive disease up to 40.51 months
Population: All participants who had at least one dose of the study drug. The numbers of participants censored are 7 (MM) and 33 (WM).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Multiple Myeloma (MM) | Waldenstrom's Macroglobulinemia (WM)
Number analyzed (Participants) | 14 | 42
months | 5.11 [2.86 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 27.73 [20.47 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

4. Secondary Outcome: Number of Participants With Adverse Events (Safety and Adverse Events)
Description: Data are presented as number of participants who experienced serious adverse events or all other nonserious adverse events during the study including the 30-day follow-up period. A summary of serious adverse events and other nonserious adverse events is located in the Reported Adverse Event section. Safety data were collected up to 24 cycles plus 30 days of follow-up for a total up to 23.40 months.
Time Frame: Treatment start to 30 days after discontinuation of study treatment up to 23.40 months
Population: All participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Multiple Myeloma (MM) | Waldenstrom's Macroglobulinemia (WM)
Number analyzed (Participants) | 14 | 42
Participants
  Serious Adverse Events | 4 | 9
  Other Nonserious Adverse Events | 12 | 42

5. Other Pre Specified Outcome: Number of Participants Who Died Due to Progressive Disease During the 30 Days Following Discontinuation From Study Treatment
Time Frame: Study treatment discontinuation up to 30 days post study treatment discontinuation
Population: All participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Multiple Myeloma (MM) | Waldenstrom's Macroglobulinemia (WM)
Number analyzed (Participants) | 14 | 42
Participants | 0 | 1

ADVERSE EVENTS:
Description: Deaths due to progressive disease are not considered adverse events; however they are reported in the Participant Flow for those who died during the study and in the Other Pre-Specified Outcome Measure for those who died during the 30-day post study treatment follow-up period.
Arm/Group | Multiple Myeloma (MM) | Waldenstrom's Macroglobulinemia (WM)
Serious Adverse Events (participants affected / at risk) | 4/14 | 9/42
Other Adverse Events (participants affected / at risk) | 12/14 | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multiple Myeloma (MM) (N=14) | Waldenstrom's Macroglobulinemia (WM) (N=42)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) — This event resulted in death.
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) — This event resulted in death within 30 days of study discontinuation.
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (2)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 (2) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) — This event resulted in death.
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Iiird nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multiple Myeloma (MM) (N=14) | Waldenstrom's Macroglobulinemia (WM) (N=42)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 14 (15)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 8 (8)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 6 (7)
Vertigo (Ear and labyrinth disorders) | 2 (6) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (9) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (11) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (2) | 2 (2)
Asthenia (General disorders) | 3 (7) | 3 (3)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 5 (7) | 22 (23)
Malaise (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 2 (4) | 1 (1)
Pyrexia (General disorders) | 4 (8) | 3 (3)
Bronchitis (Infections and infestations) | 2 (4) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 4 (5)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (3)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 9 (10)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Aphonia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 9 (9)
Head discomfort (Nervous system disorders) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 5 (6)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (2) | 2 (2)
Apathy (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 4 (11) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days